CLINICAL TRIAL: NCT06557304
Title: This is a Multicenter, Retrospective Real-world Study of BTK Inhibitor in the Treatment of Chronic Lymphocytic Leukemia in China
Brief Title: The Real World Study of BTK Inhibitor in the Treatment of Chronic Lymphocytic Leukemia in China
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Other Study IDs: BTKi-CLL-RWE
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: CLL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: BTK inhibitor — patients with treatment naive or R/R CLL who treatment with BTK inhibitor

SUMMARY:
This is a Multicenter, Retrospective Real-world Study of Zanubrutinib in the Treatment of Chronic Lymphocytic Leukemia in China

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years old
2. Must have a confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL) requiring treatment (iwCLL [International Workshop on Chronic Lymphocytic Leukemia] criteria)；
3. Treatment-naïve OR Refractory Recurrence CLL patients who were initiated on BTK inhibitor;
4. Prior or current use of BTK inhibitor for ≥3 months
5. At least one follow-up was recorded during BTK inhibitor treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators participating in this observational study should include all patients with CLL who initiated treatment with BTK inhibitor over the period from Dec. 1st, 2017 to the present, regardless of the treatment status at the time of inclusion. Thus, at the time of enrolment and retrospective data collection, patients may still be on treatment or have stopped treatment for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | up to five years
  OS is defined as the time from the starting date of BTK inhibitor to the date of death due to any cause.

SECONDARY OUTCOMES:
Time to Next Therapy (TTNT) | up to two years
  The TTNT will be calculated as the difference between BTK inhibitor initiation date and initiation date of the first next therapy for CLL
Adverse Events | up to five years
  Percentage of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Special Situations